CLINICAL TRIAL: NCT02617537
Title: A Multinational, Double-blind, Randomized, Placebo-controlled, Parallel-group Clinical Study to Investigate the Efficacy and Safety of the Oral Hormonal Contraceptive BAY 86-5300 (0.02 mg Ethinyl Estradiol as Betadex Clathrate and 3 mg Drospirenone) Over 16 Weeks for the Treatment of Women With Dysmenorrhea
Brief Title: To Investigate Efficacy of YAZ in the Treatment of Dysmenorrhea
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16419; 2015-003924-29 (EudraCT Number)
Record Dates: First submitted 2015-11-23; First posted 2015-12-01 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BAY86-5300 (Experimental): Patients suffering from dysmenorrhea, treated with Yaz
  Interventions: Drug: EE20/DRSP(YAZ,BAY86-5300)
- Placebo (Placebo Comparator): Patients suffering from dysmenorrhea,treated with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EE20/DRSP(YAZ,BAY86-5300) — 0.02 mg EE (β-CDC)/3 mg DRSP for 24 days and placebo tablets for 4 days per 28-day intake cycle
  Arms: BAY86-5300
Drug: Placebo — Matching placebo tablets for 28 days per 28-day intake cycle
  Arms: Placebo

SUMMARY:
The objective of this study is to investigate the safety and efficacy of (0.02 mg EE as betadex clathrate [β-CDC]) / 3 mg drospirenone (DRSP) for dysmenorrhea. In order to appropriately evaluate the efficacy of EE(β-CDC)/DRSP the study was set up as a placebo-controlled comparative study

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from dysmenorrhea for at least the previous 3 months prior to Visit 1 with a minimum visual analogue scale (VAS) score of 30 mm with regard to pain during the menstrual period of the screening period
* Good general health (except for findings related to dysmenorrhea) as proven by medical history
* Patients aged 18 years or older at the time of obtaining informed consent; smokers must not be older than 35 years at the time point of informed consent
* Normal or clinically insignificant cervical smear not requiring further follow up (a cervical smear has to be taken at screening visit or a normal result has to be documented within the previous six months). Human papilloma virus (HPV) testing in subjects with atypical squamous cells of undetermined significance (ASCUS) can be used as an adjunctive test. Subjects with ASCUS can be included if they are negative for high-risk HPV strains (HPV 16, HPV18).
* Women of childbearing potential must agree that adequate contraception will be used when they are sexually active. This applies from signing of the informed consent form until 2 weeks after the last study drug administration.

Exclusion Criteria:

* Pregnancy (confirmed or suspected) or lactation (less than three months since delivery, abortion, or lactation before start of treatment)
* Patients who wish to become pregnant during the course of the study
* Body Mass Index (BMI) > 32 kg/m2
* Hypersensitivity to any ingredient of the study drug
* Laboratory values outside inclusion range before randomization
* Any diseases or conditions that can compromise the function of the body systems and could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the study medication
* Any diseases or conditions that might interfere with the conduct of the study or the interpretation of the results
* Any disease or condition that may worsen under hormonal treatment according to the assessment and opinion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Mean change in visual analogue scale (VAS) score for pain due to dysmenorrhea from baseline to Visit 6 | Baseline to week 17
  The patient marks the individual pain impression on a visual analogue scale in the range 0 (no pain) to 100mm (worst pain ever experienced)

SECONDARY OUTCOMES:
Number of participants with adverse events as measure of safety and tolerability | Up to 16 weeks
Number of days with dysmenorrhea | Up to 16 weeks
  The occurrence of dysmenorrhea will be recorded in the patient diary
Change in dysmenorrhea score | Baseline to week 16
  It is the sum of two four-stage sub-scales which assess the extent to which dysmenorrhea interferes with daily life & the extent to which pain medication is used.
Changes from baseline to each menstrual period of total number of taken supportive analgesic medication | Baseline to week 16
  Standard Analgesic tablets are provided to participants
Changes from baseline to each menstrual period of days without supportive analgesic medication. | Baseline to week 16
Clinical Global Impression(CGI) | At week 16
  The CGI is the measure of global improvement index from the opinion of the investigator and subject to document changes in the health status during treatment
Self administered SF-36 questionnaire | At baseline and week 17
  The 36-items Short Form Health Survey (SF-36) (version 2.0) is a set of generic, coherent,and easily administered quality-of-life measures.
Changes from baseline to each menstrual period of severity of lumbago | Up to 16 weeks
  The patient classifies the severity on a mild, moderate, severe scale
Changes from baseline to each menstrual period of severity of headache | Up to 16 weeks
  The patient classifies the severity on a mild, moderate, severe scale
Changes from baseline to each menstrual period of severity of nausea/vomiting | Up to 16 weeks
  The patient classifies the severity on a mild, moderate, severe scale

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer